CLINICAL TRIAL: NCT05899218
Title: Sexual and Gender Minority Emerging Adults Eliciting Narratives (SEEN)
Brief Title: Sexual and Gender Minority Emerging Adults Eliciting Narratives
Acronym: SEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 853689
Record Dates: First submitted 2023-05-19; First posted 2023-06-12 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Wellness 1; Sexual Orientation; Gender Identity
Keywords: racial/ethnic identity; intersectionality; mental health treatment seeking; intervention; narrative
MeSH Terms: conditions — Sexual Behavior; Intersectional Framework; Narration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photo-Novella (Experimental): Participants in the photo-novella intervention will be asked to take 12 photographs and write a caption for each photo based on two prompts.
  Interventions: Behavioral: Critical Narrative Development
- Digital Storytelling (Experimental): Participants in the digital storytelling intervention will be asked to create two videos (1-3 minutes each) based on two prompts.
  Interventions: Behavioral: Critical Narrative Development

INTERVENTIONS:
Behavioral: Critical Narrative Development — Participants are asked to answer two prompts ("describe an experience where you have felt seen as an LGBTQ+ person of color" and "describe an experience where you have felt unseen as an LGBTQ+ person of color").

SUMMARY:
Critical narrative interventions (CNIs) have not been examined for addressing psychological outcomes (e.g., depression, anxiety, self-esteem, empowerment, psychological well-being) within sexual and gender minority emerging adults (SGM EA) of color; therefore, this pilot study will examine the use of CNIs to impact SGM of color psychological outcomes. Prior literature has shown that CNIs have the potential to increase empowerment, self-efficacy, and social support as a prevention strategy for mental health. The research study is being conducted to see if telling your story through photographs or video can improve the mental health and well-being of emerging adults that identify as a member of a sexual and/or gender minority and a racial and/or ethnic minority.

Participants will be asked to complete the following research procedures:

1. take a survey online (about 20-30 minutes), then an interview about everyday experiences as sexual/gender minority of color and your experiences in seeking out mental health services.
2. After the interview, participants will have one month to tell their story, answering two prompts "Tell us a time you have felt seen" and "Tell us a time when you have felt unseen." You will be randomized to one of two formats of telling your story: taking photographs or making two short videos.

   1. Photographs: Those that are randomized to the photograph condition will be asked to take 12 photos total telling your story and answering the prompt.
   2. Videos: Those that are randomized to the video condition will be asked to create two (1-3 minute) videos telling your story and answering the prompts.
3. At the one-month time frame, participants will be asked to fill out another survey (about 20-30 minutes) and then complete an interview about the photos or videos created.

DETAILED DESCRIPTION:
The research activities involve a two-arm pilot enrolling a sample of 30 participants who identify as sexual and gender minority (SGM), racial/ethnic minority/person of color (POC), and living with moderate to severe depression. After consent and completion of the baseline survey (15-20 min) and interview (45-60 min), participants will be randomized into one of two critical narrative interventions: photo-novella (n=15) or digital storytelling (n=15).

All participants will be given the same two prompts for their narrative intervention asking, "Share an experience of when you have felt seen as an SGM Person of Color in Philadelphia." AND "share an experience of when you have felt unseen as an SGM person of color in Philadelphia."

Photo-Novella: Participants in the photo-novella intervention will be asked to tell their story through 12 photographs and a caption (6 for the first prompt and 6 for the second prompt). Participants will be instructed to take a photograph answering the two prompts. Participants may use their smartphones or digital camera to capture their photographs. Participants may also edit their photographs using photo-editing software for aesthetics. Participants will also be asked to provide a short caption (no more than two sentences) explaining their photograph and provide a title for their work. Participants will be provided with a basic guide on photography and how to "snap a picture."

Digital Story: Participants in the digital storytelling intervention will be asked to tell their story in 3-6 minutes (two videos total, 1-3 minutes each) utilizing a video format that can include still or moving images, sound, music, and voiceover. Participants will be provided with a guide on software or applications that they can use to create their stories. Participants will be provided with a manual or basic guide to digital stories for their reference. Participants will be provided with guidance on expectations of the video, including format, length, quality, and closed captions for accessibility.

At the baseline visit after the survey and interview, participants will be randomized into one of the two intervention conditions (photo-novella or digital story). Once the participant is randomized, they will be provided with the electronic manual (based on their intervention). The research team member will provide guidance on what to expect (i.e., how many photos to take and what the prompt is) and go over the manual with the participant. The participant will then be given the opportunity to ask questions.

The participants will be given one month to complete their narrative and be asked to digitally submit their work to the research team during the 1-month visit. Participants will also be given the opportunity to present their work at a gallery (but not required to), which will be scheduled later (about ten months from the date of the first enrollment). The gallery and participation in the gallery are entirely voluntary and will not affect participation in the study.

A week before the scheduled 1-month follow-up, a research team member will reach out to the participant to confirm the 1-month study visit via phone, e-mail, or text as indicated in the participant's preferred contact method. A research team member will reach out every two days for confirmation until received from the participant.

Participants will receive a link via email a day before their one-month follow-up visit to complete a follow-up survey (15-20 mins). During the one-month follow-up, a research team member virtually on Zoom will conduct a follow-up interview (45-60 mins) asking participants about their experience of creating their critical narrative piece. At the one-month follow-up, research team members will review the final critical narratives of the participants digitally. Two days before the one-month follow-up, participants will receive a link via email to a Box folder (that is HIPAA compliant) where they can upload their photos/videos.

The participants will be notified of the gallery date and invited to attend. The gallery is optional and does not impact participation in the study.

ELIGIBILITY:
Inclusion Criteria

* identify as a sexual minority
* live in the United States
* identify as a person of color
* be aged 18-24 years
* have a smartphone and or computer access
* identify as living with moderate to severe depression as indicated on the PHQ-9 (score of 10 or higher)
* do not report suicidal ideation in the past month.

Exclusion Criteria:

* Identifies as a cisgender heterosexual man or woman
* Does not live in the United States
* Identifies as non-Hispanic white or Caucasian
* Is not between the ages of 18-24 years (inclusive)
* Does not have access to a smartphone or computer
* Plan to move out of the region for the next six months
* Does not consent to study procedures
* Meets criteria for an unmanaged psychotic disorder
* meets criteria for none to mild depression on the PHQ-9 (score of 9 or less)
* reports suicidal ideation in the past month

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tran, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- School of Nursing, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study, we plan to share with other researchers the de-identified individual participant data (IPD). This will only include the quantitative survey data collected and baseline and follow-up.
Supporting Information: Study Protocol
Time Frame: The data will be available 1 year after the completion of study. The data will be available indefiitely.
Access Criteria: Data is available for the community, academic researchers, and educational purposes.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photo-Novella | Digital Storytelling
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — deemed ineligible out of country | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photo-Novella | Digital Storytelling | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — open text box answer allowing for participants to enter in their age at time of study
  years | 20.80 (2.10) | 20.60 (1.58) | 20.70 (1.81)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex assigned a birth: Female | 8 | 8 | 16
  Sex assigned a birth: Male | 2 | 2 | 4
  Sex assigned a birth: X (third gender) | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Self-Identify as LGBTQ+ [Count of Participants; unit: Participants] — to be eligible for the study participants had to identify as a sexual or gender minority individual (LGBTQ+)
  Participants
    LGBTQ+ | 10 | 10 | 20
    non-LGBTQ+ | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: scores range from 0 to 27, higher scores indicate higher levels of depression severity.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 14.29 (4.72) | 11.50 (.93)

2. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: scores range from 0 to 21, higher scores indicate higher levels of anxiety severity.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 10.71 (5.16) | 11.00 (3.70)

3. Primary Outcome: The Flourishing Scale
Description: scores range from 8 to 56, higher scores represent an individual with many psychological resources and strengths.
Time Frame: 1 month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 39.29 (10.53) | 41.13 (6.24)

4. Primary Outcome: Rosenberg Self-Esteem Scale
Description: scores range from 8 to 56, higher scores represent an individual with higher self-esteem.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 25.43 (4.72) | 25.00 (2.98)

5. Secondary Outcome: Internalized Stigma of Mental Illness Scale (ISMI-9)
Description: scores range from 1 to 4, higher scores represent higher internalized stigma towards mental illness.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 2.64 (.23) | 2.51 (.16)

6. Secondary Outcome: LGBTQ+ POC Microaggressions Scale-Brief (LGBTQ+ PCMS-B): Racism in Dating Subscale
Description: scores range from 0 to 20 for each subscale, higher scores represent higher levels of racism in LGBT community, Heterosexism in Racial/ethnic community, and racism in dating/relationship.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 6.57 (5.50) | 2.13 (3.64)

7. Secondary Outcome: Attitudes Toward Mental Health Treatment (ATMHT) Scale
Description: scores range from 20 to 80, higher scores represent more positive attitudes towards mental health treatment seeking.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 57.86 (9.41) | 45.63 (13.26)

8. Secondary Outcome: General Belongingness Scale (GBS): Sense of Acceptance Sub Scale
Description: scores range from 12 to 84, higher scores represent higher sense of belonging.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 24.57 (6.16) | 23.75 (6.25)

9. Secondary Outcome: Multidimensional Scale of Perceived Social Support (MSPSS)
Description: scores range from 1 to 7, higher scores represent higher perceived social support.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 5.69 (.96) | 4.69 (.93)

10. Secondary Outcome: Intersectional Discrimination Index -Anticipated Discrimination (InDI-A)
Description: scores range from 0 to 4, higher scores represent higher anticipated intersectional discrimination
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 2.17 (.73) | 2.47 (.79)

11. Secondary Outcome: The Queer People of Color Identity Affirmation Scale (QPIAS): Identity Based Growth Subscale
Description: two subscales, identity based growth with scores from 7 to 49 with higher scores representing higher growth, and identity cohesion with scores from 5 to 35 with higher scores as higher identity cohesion
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 35.57 (11.69) | 32.88 (5.79)

12. Other Pre Specified Outcome: Acceptability of the Intervention Measure (AIM)
Description: scores range from 5 to 20, higher scores represent higher acceptability for the intervention.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 18.43 (2.30) | 16.25 (3.58)

13. Other Pre Specified Outcome: Intervention Appropriateness of the Measure (IAM)
Description: scores range from 5 to 20, higher scores represent higher appropriateness of the intervention.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 18.71 (2.21) | 16.37 (2.07)

14. Other Pre Specified Outcome: Feasibility of the Intervention Measure (FIM)
Description: scores range from 5 to 20, higher scores represent higher feasibility for the intervention
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photo-Novella | Digital Storytelling
Number analyzed (Participants) | 7 | 8
score on a scale | 16.86 (2.79) | 16.38 (2.88)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 1 month during participants enrollment in the study
Arm/Group | Photo-Novella | Digital Storytelling
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05899218/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT05899218/ICF_001.pdf